CLINICAL TRIAL: NCT00003256
Title: A Phase II Trial of Flavopiridol in Patients With Metastatic Androgen Independent Prostate Cancer
Brief Title: Flavopiridol in Treating Patients With Recurrent Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000066145; WCCC-CO-9781; NCI-T97-0038
Record Dates: First submitted 1999-11-01; First posted 2004-08-02 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2013-01

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage IV prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — alvocidib

ARMS (1):
- Arm I (Experimental): Patients receive intravenous flavopiridol over 72 hours every 2 weeks for at least 4 courses. After 2 courses of treatment, patients not experiencing unacceptable toxic effects may receive a dose escalation.
  Interventions: Drug: alvocidib

INTERVENTIONS:
Drug: alvocidib

SUMMARY:
Phase II trial to study the effectiveness of flavopiridol in treating patients with recurrent prostate cancer after hormone therapy. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Evaluate the clinical effectiveness of flavopiridol in patients with metastatic androgen independent adenocarcinoma of the prostate.

II. Assess the toxic effects of flavopiridol in this patient population.

OUTLINE:

Patients receive intravenous flavopiridol over 72 hours every 2 weeks for at least 4 courses. After 2 courses of treatment, patients not experiencing unacceptable toxic effects may receive a dose escalation. Patients are followed every 3 months until death.

ELIGIBILITY:
PATIENT CHARACTERISTICS:

* Performance Status: ECOG 0-2
* Life Expectancy: At least 3 months
* WBC at least 3,000/mm3
* Absolute neutrophil count at least 1,200/mm3
* Platelet count at least 100,000/mm3
* Hemoglobin at least 8 g/dL
* Bilirubin no greater than 1.5 mg/dL
* SGOT no greater than 2.5 times normal
* Creatinine no greater than 1.5 mg/dL
* Prostate-specific antigen at least 10 ng/mL (if bone only disease)
* No prior or concurrent maligancies within 5 years, except nonmelanoma skin cancer
* No serious medical illness
* No cord compression symptoms

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy
* No prior suramin therapy
* Prior or concurrent use of luteinizing hormone-releasing hormone allowed (no other concurrent hormonal therapy)
* No prior anti-androgen therapy within 4 weeks of study
* At least 4 weeks since prior radiotherapy
* No prior strontium therapy

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 1998-05; Primary Completion 2002-07 (Actual); Study Completion 2004-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Wilding, MD, Study Chair — University of Wisconsin, Madison
Locations (4):
- United States (4):
  - Beckman Research Institute, City of Hope, Duarte, California
  - University of California Davis Cancer Center, Sacramento, California
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin

REFERENCES:
- [Result] Liu G, Gandara DR, Lara PN Jr, Raghavan D, Doroshow JH, Twardowski P, Kantoff P, Oh W, Kim K, Wilding G. A Phase II trial of flavopiridol (NSC #649890) in patients with previously untreated metastatic androgen-independent prostate cancer. Clin Cancer Res. 2004 Feb 1;10(3):924-8. doi: 10.1158/1078-0432.ccr-03-0050. PMID 14871968